



## Polyvagal Informed Group Skills Training for Body Awareness and Managing Emotions for People Living with Obesity

**Informed Consent Form** 

19th of October 2025





## **Informed Consent Form**

Study Title: Group polyvagal theory informed therapy for body awareness and managing emotions for people living with obesity

| Tick here: |
|---|
| The nature and purpose and potential benefits or risks of the study have been explained to me. I have watched the information video read and understood the participant information sheet (version 4) and understand what this study involves. If I asked questions, they have been answered fully to my satisfaction. |
| I can commit for up to 16 weeks for the entirety of the study and understand the commitment needed in terms of completing daily and weekly online questionnaires on the platform Qualtrics. |
| I agree to the video and audio recording of the group sessions on Microsoft Teams for the purpose of clinical supervision and to help ensure the group is delivered effectively. I understand that the recordings will only be accessed by the research team, and will not be used for any other purpose. I understand that the recordings will be stored on an NHS Microsoft SharePoint account, which is a Trust-approved encrypted platform and is password protected, for a maximum of 9 weeks, after which they will be destroyed. |
| I understand that my participation in the study is entirely voluntary and that I am free to withdraw at any time without giving a reason. |





| I agree that if I decide to withdraw from the study then the researchers can continue to use the data and information I have already given them unless I ask for this to be destroyed. |
|---|
| Agree to my GP being informed that I'm taking part in the study. |
| I understand that all data will be kept confidential and that no personal, identifying information will be disclosed in any reports on the project, or to any other party. |
| I understand that the researcher may contact my care team, GP or relevant authorities if they are concerned about my safety or the safety of others. |
| I agree to take part in the study. |
| Participant signature: Date: |